CLINICAL TRIAL: NCT04161911
Title: Overall Survival and Treatment Patterns for Advanced Hepatocellular Carcinoma Patients Who Received Second or Third Line Nivolumab Therapy
Brief Title: A Study to Assess Overall Survival and Treatment Patterns for Advanced Liver Cancer Participants Who Received Nivolumab Therapy
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-79L
Record Dates: First submitted 2019-11-12; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Hepatocellular Carcinoma (aHCC) cohort: aHCC cohort selected from the Flatiron Health Oncology electronic health record (EHR) data from January 2011 to the most recent data available. The index date will be defined as the start of second or third line nivolumab therapy for aHCC between January 1, 2011 and the most recent data available.

SUMMARY:
A study to describe real-world treatment patterns and overall survival in advanced liver cancer participants who received second or third line nivolumab therapy

DETAILED DESCRIPTION:
The central aims of this study are descriptive and designed to describe the patient demographics, clinical characteristics, treatment patterns, and overall survival in advanced liver cancer participants who received second or third line nivolumab therapy in the real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult aHCC participants in the Flatiron database as defined by:
* Diagnosed with HCC International Classification of Diseases (ICD)-9 155.x or ICD-10 C22.x)
* Pathology consistent with advanced HCC
* Age 18 years or older at index
* At least two clinic encounters on different days in the Flatiron database occurring on or after January 1, 2011
* Participants who received second or third line nivolumab monotherapy or combination therapy for aHCC

Exclusion Criteria:

* Participants with <1 month of medical data (any clinic visits, medication administrations or oral medication prescriptions) following and including the index date
* Participants with clinical study drug during prior or post study index periods

Other protocol-defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will be selected from the Flatiron database according to the inclusion and exclusion criteria.
  Participants will be eligible for inclusion in this study if:
  1. Diagnosed with advanced Hepatocellular Carcinoma (aHCC) in the Flatiron database;
  2. Aged 18 years or older at index date; and
  3. Received second or third line nivolumab monotherapy or combination therapy for aHCC.
  Participants will be excluded if:
  1. Received clinical study drugs prior to, on, or post the index date;
  2. Have less than 1 month of medical data following and including the index date. Those meeting the inclusion and exclusion criteria will be further stratified by lines of therapy and Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score.
Sampling Method: Probability Sample
Enrollment: 1426 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Treatment patterns | From aHCC diagnosis date to first nivolumab treatment (Up to 7.75 years)
  Nivolumab second and third lines of therapy will be described including prior lines of therapy, duration of nivolumab therapy and time from aHCC diagnosis date to first nivolumab treatment
Overall Survival | From start date of 2L and 3L nivolumab therapy to the date of death (Up to 7.75 years)
  The initial second or third line nivolumab therapy date will be used as the start date for the OS analysis. Occurrence of death will be considered as event and the duration for event will be calculated as time from 2L or 3L nivolumab therapy date to death date. Patients who survived will be censored and their duration period will be the time between the initial 2L or 3L nivolumab therapy date and the last date of their post-period follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol Myers Squibb, CORDS Research, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm